CLINICAL TRIAL: NCT06618131
Title: Examination of the Effects of Virtual Reality Exercises on Lower Extremity Skin Temperature, Arterial Stiffness, Gait Parameters and Enjoyment of Exercise in Individuals With Peripheral Arterial Disease
Brief Title: Effects of Virtual Reality Exercises on Individuals With Peripheral Artery Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ayten Demir, Graduate Student, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEU-FTR-AE-01
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Arterial Disease(PAD)
Keywords: virtual reality; exercise; arterial stiffness; gait analysis; skin temperature
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercising with Virtual Reality (Active Comparator): 12 participants will undergo a virtual reality exercise program with the X-Box 360 KinectTM game console (X-Box 360, Microsoft, United States of America) for 50 minutes a day, 2 days a week for 12 weeks.
  Interventions: Other: Exercise
- Control Group (No Intervention): In this group of 12 people, there will be no intervention.

INTERVENTIONS:
Other: Exercise — Exercise program with virtual reality applications for lower extremities
  Arms: Exercising with Virtual Reality

SUMMARY:
The aim of this study is to investigate the effects of virtual reality exercises on lower extremity skin temperature, arterial stiffness, gait parameters and enjoyment of exercise in individuals with peripheral arterial disease.

DETAILED DESCRIPTION:
The number of studies conducted in individuals with peripheral arterial disease (PAD) is quite small. In the only existing study, it was found that the application of a walking program on a treadmill in a virtual environment created with virtual reality increased the walking distance of individuals with intermittent claudication. In this direction, our study was planned to determine the effect of exercise program with virtual reality application on skin temperature, arterial stiffness, gait parameters and exercise enjoyment in individuals with PAD.

The study group will receive an exercise program with X-Box 360 KinectTM game console (X-Box 360, Microsoft, United States) for 50 minutes a day, 2 days a week for 12 weeks, and the control group will receive only a home exercise program. Lower extremity skin temperature will be evaluated with a thermal camera (FLIR E53, FLIR Systems, Wilsonville, Oregon, USA), arterial stiffness will be evaluated with an arterial stiffness meter (SphygmocorXCEL device), gait parameters will be evaluated with a wearable movement analysis system (G-walk), 6 Minute Walk Test and Walking Impairment Questionnaire. Enjoyment of physical activity will be evaluated with The Short Version of Physical Activity Enjoyment Scale Assessments will be made as initial assessment before the exercise program, interim assessment at week 6 and final assessment at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with PAD
* Being between 18-65 years of age
* Ankle-brachial index less than 0.9
* Not having a lower extremity injury or surgery that would prevent participation in the exercise program

Exclusion Criteria:

* History of cardiovascular events less than 3 months before the start of the study
* Uncontrolled severe hypertension (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg)
* Uncontrolled diabetes mellitus (glycemic index ≥ 290)
* Critical Limb Ischemia
* Balance Problems
* Vertigo
* History of epilepsy
* Dementia
* Chronic diseases that may be contraindications for exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Skin Temperature, | Twelve weeks
  In our study, a thermal camera (FLIR E53, FLIR Systems, Wilsonville, Oregon, USA) with a temperature sensitivity of 0.04°C will be used to record lower extremity skin temperature with real-time imaging.Controls related to thermographic scaling will be performed according to Thermographic Imaging in Sports and Exercise Medicine (TISEM)" criteria.

SECONDARY OUTCOMES:
Arterial Stiffness Measurement | Twelve weeks
  Arterial stiffness represents the viscoelastic properties of the vessel wall, indicates vascular damage and is a measure of the degree of atherosclerosis. Increased arterial stiffness or decreased compliance is indicative of extensive atherosclerotic involvement of the vasculature. One of the non-invasive techniques used to assess arterial stiffness is pulse wave analysis (PWA). PWA examines pressure waveforms within the main arteries. Pulse wave velocity (PWV) and enhancement index (Alx) are indices of arterial stiffness.PWV is the velocity of the pulse propagating along the arterial segment. Alx is the ratio of the difference between the late systolic pressure reflected from the periphery and the early systolic pressure to the pulse pressure, expressed as a percentage. The SphygmoCor XCEL device will be used to assess arterial stiffness.
Wearable Motion Analysis System | Twelve weeks
  The dynamic gait parameter will be assessed with the BTS G-Walk Device, a wearable movement analysis system. The BTS G-Walk sensor system is a wireless magnetic sensor device that can be used to determine spatio-temporal parameters as well as pelvic movements during walking. The system consists of many parameters that analyze movements such as walking, running and jumping. In gait analysis, this system compares bilateral right and left limbs with normal values, and provides kinematic analysis of the pelvis in 3 planes.
Six-Minute Walk Test | Twelve weeks
  The test will be performed along a 30 meter long by 1.5 meter wide corridor according to standard procedures developed by the American Thoracic Society. Participants will be instructed to walk along the 30-meter corridor from the starting point to the end at the best speed they can within 6 minutes, using standard encouragement phrases at the beginning of each minute. Modified Borg Scale will be used for dyspnea and leg fatigue perception. At the end of the test, the total distance covered will be recorded in meters (m). The calculation of percentage values will be based on the reference values formulated by Enright et al. in healthy population.
Walking Impairment Questionnaire (WIQ) | Twelve weeks
  To assess intermittent claudication, the Turkish adaptation of the 21-item self-report scale Decreased Walking Distance Scale developed by Dr. Regensteiner et al. (1995) will be used. The scale consists of claudication, differential diagnosis, distance, speed and stair parameters. The sub-parameters (distance, speed and stairs) are rated on a Likert scale ranging from 0 (unable, very difficult) to 4 (no difficulty at all) and each item has a weighted score. The claudication and differential diagnosis section is assessed individually, while the subscales are assessed on a scale of 0 to 100 points, calculated according to the weight of each question. The subscale score is obtained by dividing the Likert scale score by the maximum weighted score and multiplying by 100. Each subscale score is evaluated between 0-100. A high score indicates high performance. Total and combined scores are calculated by averaging the subscales.
Short Version of Physical Activity Enjoyment Scale | Twelve weeks
  The physical activity enjoyment scale is an 18-item scale developed to assess the enjoyment of physical activity in young adults (Kendzierski & DeCarlo, 1991). The short form of the physical activity enjoyment scale (8 questions) was adapted from the original 18-item scale by Raedeke. The Turkish validity and reliability of the scale was conducted by Soylu et al. The Exercise Enjoyment Scale consists of 8 items with a 7-point Likert-type rating and a single dimension. The scale evaluates positive emotions such as enjoyment and pleasure from exercise. A high mean score on the scale indicates that the level of enjoyment from exercise is high, while a low mean score on the scale indicates that the level of enjoyment from exercise is low.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Faculty of Physical Therapy and Rehabilitation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The reason for not sharing data is the concern about unauthorized use.